CLINICAL TRIAL: NCT00867204
Title: Prospective Randomized Blinded Comparison of a Short-wire ERCP System to Traditional Long-wire Devices
Brief Title: Short Versus Long Wire ERCP Systems
Acronym: ERCP systems
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: ERCP systems
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2009-03

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography
Keywords: ERCP; Study focus was to compare the performance of the ERCP short-wire device versus the Long-wire device.
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Short-wire device: The Fusion Short-wire ERCP device was used
  Interventions: Procedure: ERCP
- Long-wire device: The traditional Long-wire ERCP device was used
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — Patients with clinical indication for ERCP were invited to participate in the Study

SUMMARY:
This study looked at short-wire ERCP devices versus Long-wire ERCP devices. The study hypothesis is to compare the performance of the Fusion ERCP short-wire system to the traditional Long-wire system.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing ERCP.

Exclusion Criteria:

* Age less than 18 years, pregnant women, patients unable to provide informed concent, prior surgery causing a significant change in the anatomy of the papilla (Billroth II or Roux-en-Y)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with the clinical indication for an ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2004-10; Primary Completion 2008-02 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Time for device exchange and stent insertion | during the ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Draganov, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida/Shands UF Endoscopy Center, Gainesville, Florida, United States